CLINICAL TRIAL: NCT05585463
Title: Safety of Acupuncture and Intracutaneous Needles in Pediatric Cancer Patients: a Retrospective Study
Brief Title: Safety of Acupuncture and Intracutaneous Needles in Pediatric Cancer Patients: a Retrospective Study (ACUSAFE2021)
Acronym: ACUSAFE2021
Status: Completed | Type: Observational
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Principal Investigator, Esther Martinez Garcia, Head of integrative pediatric oncology. Pediatric Cancer Center Barcelona, Hospital Sant Joan de Deu, Fundació Sant Joan de Déu
Other Study IDs: PS-14-22
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Cancer Pediatric; Neutropenia; Thrombocytopenia; Bacteremia; Infection;Skin;Localised; Safety Issues
Keywords: Acupuncture; Intracutaneous Needle; Cancer; Children; Neutropenia; Thrombocytopenia; Infection; Safety; Bacteremia
MeSH Terms: conditions — Neoplasms; Neutropenia; Thrombocytopenia; Bacteremia; Infections | interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Oncology pediatric patients treated with acupuncture: Patients in the oncology area of the Sant Joan de Déu Hospital treated at the UOPI (Integrative Pediatric Oncology Unit) from September 2019 to September 2021 have received treatment with acupuncture and intracutaneous Seirin New Pyonex Press Tack®.
  Patients in active treatment and survivors are included. Acupuncture treatment can be received in a hospitalization ward, an intensive care unit, a day hospital or an outpatient clinic.
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — Acupuncture with needles and intracutaneous needles in the ear or body. The insertion is done with gloves, a guide to puncture the needle, and exhaustive skin disinfection.

SUMMARY:
This study aims to demonstrate the safety of intracutaneous needles in pediatric cancer patients. For this, a two-year retrospective study will be carried out to determine the incidence of adverse effects related to acupuncture and the use of intracutaneous needles in the patient in active treatment and survivor.

DETAILED DESCRIPTION:
Retrospective study of review of medical records. It is a single-center, descriptive, observational study. There are no comparison or control groups. No type of patient selection (randomization or blinding) will be performed.

The medical records of patients treated at the Integrative Pediatric Oncology Unit from September 2019 to September 2021 who have received acupuncture treatment (disposable intracutaneous needles) will be reviewed.

The number of treatments applied, the localization of the treatment, the average number of sessions per patient, and the total number of intracutaneous needles and punctured needles from September 2019 to September 2021. Likewise, the blood cultures and other adverse effects will be reviewed up to 72 hours after the removal of the needles and the intracutaneous needles (Seirin New Pyonex Press Tack®).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric oncology patients from September 2019 to September 2021 who have received treatment with acupuncture.
* Pediatric oncology patients from September 2019 to September 2021 who have received treatment with intracutaneous needles (Pyonex).

Exclusion Criteria:

* Pediatric oncology patients who have not received treatment with acupuncture or intracutaneous needles.

Ages: 1 Day to 34 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients diagnosed with developmental cancer who have been treated with acupuncture and intracutaneous needles in the Integrative Pediatric Oncology Unit of the Sant Joan de Deu Hospital in Barcelona, Spain. Such patients include patients in active treatment and survivors.
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of local infection | From the first day of needle insertion to the fourth day (withdrawal of the intracutaneous needle)
  To calculate the incidence of local infection in pediatric oncology patients during the days that the intracutaneous Seirin New Pyonex Press Tack® needles have been inserted.
  The result can be "yes" or "no".
Incidence of bacteremia | 72 hours after removal intracutaneous needle
  Analyze the incidence of positive blood cultures for gram-positive cocci up to 72 hours after removal of the intracutaneous Seirin New Pyonex Press Tack® needles.
  The result can be "yes" or "no".

SECONDARY OUTCOMES:
Incidence of bruising or bleeding | From the first day of needle insertion to the fourth day (withdrawal of the intracutaneous needle)
  To calculate the incidence of bruising or bleeding in pediatric oncology patients during the days that the intracutaneous Seirin New Pyonex Press Tack® needles have been inserted.
  The result can be "yes" or "no".
Incidence of sepsis | From the first day of needle insertion to the fourth day (withdrawal of the intracutaneous needle)
  To analyze the incidence of sepsis due to gram-positive cocci up to 72 hours after the removal of the intracutaneous Seirin New Pyonex Press Tack® needles.
  The result can be "yes" or "no".
Incidence of skin erosion | From the first day of needle insertion to the fourth day (withdrawal of the intracutaneous needle)
  Identify other skin erosion related to acupuncture and its related techniques. The result can be "yes" or "no".
Number of acupuncture needles | The day of the application of the acupuncture treatment
  Count the number of needles inserted on the day of the event (treatment The result is a minimum of one needle. This data is recorded in all acupuncture interventions and can be consulted in the clinical history.
Number of intracutaneous needles | The day of the application of the acupuncture treatment
  Count the number of intracutaneous needles inserted on the day of the event (treatment The result is a minimum of one needle. This data is recorded in all acupuncture interventions and can be consulted in the clinical history.
Degree of neutropenia | The day of the application of the acupuncture treatment in patients in oncological treatment. In survivors, the last available, up 365 days
  Report the patient's absolute neutrophil count and degree of neutropenia on the day of receiving acupuncture treatment (needles and/or Seirin New Pyonex Press Tack®).
  The Common Terminology Criteria for Adverse Events (CTCAE) is widely accepted as the standard classification and severity grading scale for adverse events in cancer therapy, clinical trials, and other oncology settings will be used. The lowest degree is 1 and the maximum is 5
Degree of thrombocytopenia | The day of the application of the acupuncture treatment in patients in oncological treatment. In survivors, the last available, up 365 days
  Report the patient's absolute platelets count and degree of thrombocytopenia on the day receiving acupuncture treatment (needles and/or Seirin New Pyonex Press Tack®).
  The Common Terminology Criteria for Adverse Events (CTCAE) is widely accepted as the standard classification and severity grading scale for adverse events in cancer therapy, clinical trials and other oncology settings will be used. The lowest degree is 1 and the maximum, 5
Type of acupuncture treatment | The day of the application of the acupuncture treatment
  • Report whether the applied treatment has been auricular (insertion of Seirin New Pyonex Press Tack® in the auricular pavilion), corporal or mixed (both techniques are performed).
  This data is recorded in all acupuncture interventions and can be consulted in the clinical history.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Martínez García, MD, Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona, Spain